CLINICAL TRIAL: NCT06937411
Title: A Phase I, Randomized, Double-Blinded, Placebo-Controlled, 2-Part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending and Multiple Ascending Doses of DC-853 in Healthy Participants
Brief Title: A Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of DC-853 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 18880; J5C-MC-FOAD (Other: Eli Lilly and Company); 2022-003220-40 (EudraCT Number)
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY4100511 (DC-853) Part 1 (Experimental): Single doses of LY4100511 (DC-853) administered orally.
  Interventions: Drug: LY4100511
- LY4100511 (DC-853) Part 2 (Experimental): Multiple doses of LY4100511 (DC-853) administered orally.
  Interventions: Drug: LY4100511

INTERVENTIONS:
Drug: LY4100511 — Administered orally
  Other Names: DC-853

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of LY4100511 (DC-853) after single and multiple dose administrations in healthy participants.

Participation could last up to 7 weeks

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to understand and comply with the requirements of the study, as judged by the Investigator.
* Participants must have a body mass index (BMI) ≥ 18 and ≤ 35 kilograms per meter squared (kg/m2).

Exclusion Criteria:

* History or presence of any clinically relevant acute or chronic medical or psychiatric condition that could interfere with the participant's safety during the clinical study or expose the participant to undue risk as judged by the Investigator.
* Malignancy within the past 5 years of screening with the exception of in situ removal of basal cell carcinoma, resected benign colonic polyps, or adequately treated cervix carcinoma in-situ.
* Planned major surgery within duration of the study or the 30 days following study completion.
* Females who are pregnant, breast feeding, lactating or plan to be pregnant during the study period or 90 days after.
* History of any drug and/or alcohol abuse in the past 2 years prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) Part 1 | Baseline up to 6 Days
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) Part 2 | Baseline up to 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- The Medicines Evaluation Unit Ltd., Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No